CLINICAL TRIAL: NCT05914428
Title: Biomarkers to Predict Acute Respiratory Distress Syndrome(ARDS) in Patients With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020BIPROSALDH2
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Sepsis
Keywords: sepsis; ARDS
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sepsis: We selected blood samples from sepsis patients from the biological bank of Qilu hospital.The ALDH2 genotype (rs671) was detected in these septic patients and divided into ALDH2 wild-type ,ALDH2 rs671 mutation.
  Interventions: Other: ALDH2 rs671 mutation

INTERVENTIONS:
Other: ALDH2 rs671 mutation — We selected blood samples from sepsis patients from the biological bank of Qilu hospital and tested their genotypes. The intervention group was ALDH2 rs671 mutation patients

SUMMARY:
Sepsis-induced acute respiratory distress syndrome (ARDS) is a life-threatening acute inflammatory lung injury, associated with increased pulmonary microvascular permeability, increased lung weight, and loss of aerated lung tissue.Despite advances in critical care, no established and targeted treatment for ARDS, contributing to a persistently high mortality rate of 34% to 45%. Therefore, exploring novel therapeutic targets for septic ARDS is of paramount importance.Acetaldehyde dehydrogenase 2 (ALDH2) is a mitochondrial enzyme that serves as the primary toxic aldehyde scavenger and is expressed in various cells, including neutrophils. The ALDH2 rs671 single nucleotide polymorphism, leading to an approximate 90% decrease in ALDH2 enzymatic activity, is implicated in occurrence of macrovascular conditions, such as coronary artery disease, pulmonary arterial hypertension, and aortic aneurysm or dissection.An array of studies has delved into role of ALDH2 in regulating cellular processes, including inflammation, autophagy, apoptosis, necrosis,efferocytosis and pyroptosis.but whether it associated with the incidence of septic-ARDS remains unknown.The aim of this study was to determine whether the ALDH2 rs671 single nucleotide polymorphism was associated with the incidence of septic-ARDS.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the ICU who were aged 18 to 85 years with a diagnosis of sepsis.Sepsis was assessed according to the third international consensus definition as life-threatening organ dysfunction caused by a dysregulated host response to infection; organ dysfunction was defined as an acute change in total Sequential Organ Failure Assessment (SOFA) score of ≥2 points consequent to the infection.

Exclusion Criteria:

1. interstitial lung disease, chronic obstructive pulmonary disease or congestive heart failure;
2. nerve injury or disease with likely prolonged ventilation；
3. the use of long-term oxygen therapy or noninvasive ventilation at home;
4. pregnancy or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conducted a single-centre, retrospective cohort study of patients diagnosed with sepsis, consecutively admitted to the intensive care unit of Qilu Hospital,Shandong university during 2020.9-2022.3,except for holidays.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Temporal dynamics of PaO2/FiO2 | From ICU administration to days 7
  PaO2/FiO2 or SpO2 / FiO2 was recorded on ICU admission，day 1 and 7
Progression to ARDS within 7 days (Berlin criteria) | From ICU administration to days 7
  The proportion of patients with sepsis progressing to ARDS

SECONDARY OUTCOMES:
Mechanical ventilation days | From administration to discharge hospital, up to 90 days
  Days of mechanical ventilation from study drug administration to discharge of ICU
Length of hospital stay | From administration to discharge hospital, up to 90 days
  The number of days the subject stayed in the hospital
Length of ICU stay | From administration to discharge ICU, up to 90 days
  The number of days the subject stayed in the ICU
incidence of septic shock | From administration to discharge ICU, up to 90 days
  incidence of septic shock

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China